CLINICAL TRIAL: NCT01729390
Title: Varying the Energy Density and Portion Size of the Main Course After a First-course Salad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutritional Sciences and Director of the Laboratory for the Study of Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FoodED501; 5R01DK059853-11 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: Feeding behavior
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Std ED Control (Experimental): 100% energy density and 133% portion size
  Interventions: Other: Energy density and portion size feeding study
- Inc ED Control (Experimental): 133% energy density and 133% portion size
  Interventions: Other: Energy density and portion size feeding study
- Std ED and Std PS (Experimental): 100% energy density and 100% portion size
  Interventions: Other: Energy density and portion size feeding study
- Std ED and Inc PS (Experimental): 100% energy density and 133% portion size
  Interventions: Other: Energy density and portion size feeding study
- Inc ED and Inc PS (Experimental): 133% energy density and 133% portion size
  Interventions: Other: Energy density and portion size feeding study
- Inc ED and Std PS (Experimental): 133% energy density and 100% portion size
  Interventions: Other: Energy density and portion size feeding study

INTERVENTIONS:
Other: Energy density and portion size feeding study — In a crossover design, adults are served breakfast and lunch, 1 day a week for 6 weeks. Breakfast is not varied across weeks. At 4 of the lunch meals, a salad first course will be served that needs to be eaten in its entirety. At these 4 meals the lunch entree will vary in energy density (100% and 133%) and portion size (100% and 133%). At the 2 lunch meals for which no first course is served, the lunch entree will be vary in energy density (100% and 133%) but be the same portion size (133%).

SUMMARY:
The purpose of this research is to determine whether varying the energy density and portion size of the main course will affect meal energy intake after consumption of a first course that has previously been shown to enhance satiety. It is hypothesized that increasing either the energy density or portion size of the main course will increase meal energy intake after consumption of the first course. It is also hypothesized that compared to when a first course is consumed, not consuming a first course will increase meal energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Adults from Penn State and the surrounding community

Exclusion Criteria:

* Currently dieting
* Food allergies

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Energy intake | 6 weeks

SECONDARY OUTCOMES:
Food intake | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States